CLINICAL TRIAL: NCT07032896
Title: 'The Effect of Nurse-Led Education on Patients' Self-Care Behaviour, Self-Efficacy Level, Medication and Diet Compliance in Individuals With Heart Failure'.
Brief Title: The Effect of Nurse-Led Education in Heart Failure Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Şengül Akdeniz, Assistant Professor , PhD, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AU-IMN-SA-01
Record Dates: First submitted 2025-05-26; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Heart Failure
Keywords: Nursing; self-care; Nursing education; Nursing care
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: The research is a randomized controlled experimental study.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): The experimental group will be trained. The training program will be implemented in line with the patient needs determined by the researcher. In order to fill this knowledge gap, existing research findings and evidence-based treatment guidelines have been extensively reviewed. The training program will be based on the guidelines. Before the patient is discharged, the patients who will be included in the intervention group will be interviewed and their verbal and written consents regarding participation in the study and application of the study forms will be obtained. The intervention group will be evaluated at the beginning of the study before training is provided and at the end of the third month when all training sessions are completed.
  Interventions: Behavioral: Nurse-led Patient Education
- Control group (No Intervention): control group routine care

INTERVENTIONS:
Behavioral: Nurse-led Patient Education — The training program will be implemented in line with patient needs determined by the researcher. In order to overcome this lack of information, existing research findings and evidence-based treatment guidelines were extensively reviewed. The training program will be based on the following guidelines. The program will start with a 30-minute individual training session on patients' self-efficacy level, self-care behaviors, medication and diet compliance processes. This training will be carried out in the hospital in accordance with the patient's plan. Discharged intervention group patients will then be interviewed by telephone six times over a period of three months, and two interviews will be scheduled for each of these monthly periods. In order to measure the impact of the intervention, data will be collected twice, before and after the training for the intervention group
  Arms: intervention group

SUMMARY:
The aim of this study is to evaluate the effect of nurse-led education on patients' self-efficacy levels, self-care behaviors, medication compliance, and diet compliance in individuals diagnosed with heart failure. This study will be conducted as a randomized controlled experimental study.

DETAILED DESCRIPTION:
This study, to be conducted at the Akdeniz University Hospital Cardiology Department and Outpatient Clinic, aims to evaluate the impact of nurse-led education on heart failure patients' self-efficacy, self-care behaviors, and adherence to medication and diet.

Study Population The study sample will comprise heart failure patients aged 18 years and older who are followed in the Cardiology Clinic at Akdeniz University Hospital.

Data Collection Instruments

The following data collection tools will be used in the study:

Patient Information Form: To collect demographic and clinical information. European Heart Failure Self-Care Behavior Scale-12: To assess self-care behaviors specific to heart failure.

General Self-Efficacy Scale: To measure perceived competence in coping with general difficulties.

Beliefs about Medication Adherence Scale: To evaluate patients' beliefs regarding adherence to medication.

Beliefs about Dietary Adherence Scale: To assess patients' beliefs concerning adherence to dietary recommendations.

Permissions for the use of the Turkish adaptations of these scales have been obtained via email from the authors responsible for their respective adaptations.

Intervention Program and Control Group An educational booklet, developed by the researcher based on a review of current research and evidence-based treatment guidelines, will be utilized for the training program, considering the specific needs of the patients.

Intervention Group: Patients in this group will receive a comprehensive educational program:

In-Hospital Individual Training: This will begin with a personalized training session conducted in the hospital, tailored to each patient's unique needs. The content of this session, covering self-efficacy, self-care, and medication and diet compliance, has been developed from an extensive review of up-to-date research and evidence-based treatment guidelines to ensure its effectiveness.

Post-Discharge Telephone Follow-up: After discharge, patients in the intervention group will receive six telephone calls over a three-month period, with two calls scheduled each month. These calls will help reinforce the in-hospital education and provide continuous support.

Control Group: This group will continue to receive routine nursing care and treatment in the Cardiology Clinic, without any additional educational interventions.

Data Collection Schedule

To measure the impact of the intervention, data will be collected twice for both groups:

Baseline: Data will be collected at the beginning of the study. Three Months Later: A second round of data collection will be conducted three months after the initial data collection.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have been diagnosed with heart failure in the hospital by a specialist physician,
* Have stable class I-IV heart failure according to the New York Heart Association (NYHA) classification criteria,
* Literate,
* Patients whose clinical condition has stabilized,
* Diabetes and hypertension under control,
* Age 18 and over,
* Have acute and chronic heart failure
* Individuals who accept the study will be included in the study.

Exclusion Criteria:

* Those with a neuromuscular problem,
* Those with serious cognitive problems and psychiatric illnesses,
* Those with physical limitations (such as visual or hearing impairment, orthopedic problems),
* Those under the age of 18,
* Those who are illiterate,
* Those who wish to withdraw from the study at any stage of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
European Heart Failure Self-Care Behaviour Scale (EHFScBS) | This assessment will be conducted at two distinct time points: at the beginning of the study (baseline- day 0) and at the end of the 3rd month.
  The European Heart Failure Self-Care Behavior Scale consists of 12 questions related to life activities to assess the self-care of Heart Failure patients. The scale is a five-point Likert-type scale with a maximum score of 60 and a minimum score of 12. Higher scores on the scale indicate better self-care behavior.The European Heart Failure Self-Care Behavior Scale (EHFScBS) will be utilized to assess changes in patients' self-care behavior levels. This longitudinal approach will allow researchers to observe any improvements or changes in self-care behaviors that may be attributable to the intervention (nurse-led in-hospital education and post-discharge telephone follow-up).

SECONDARY OUTCOMES:
General Self-Efficacy (GSE), The Beliefs About Medication Compliance Scale (BMCS), The Beliefs About Dietary Compliance Scale (BDCS) | This assessment will be conducted at two distinct time points: at the beginning of the study (baseline- day 0) and at the end of the 3rd month.
  General Self-Efficacy Scale This scale is designed to assess an individual's perceived competence in dealing with general life difficulties. It's a 4-point Likert-type scale. Scores range from a minimum of 10 to a maximum of 40. A higher score on this scale indicates that the individual has a stronger perception of their own competence.
  Beliefs About Diet and Medication Adherence Scales Both the Beliefs About Diet Adherence Scale and the Beliefs About Medication Adherence Scale are used to understand patients' beliefs regarding their adherence to dietary recommendations and medication regimens, respectively. Each of these scales comprises 12 items and uses a 5-point Likert-type scale.The minimum score on these scales is 12 and the maximum score is 60.
  Higher scores on these scales indicate that the individual has stronger beliefs about adherence to diet or medication. Conversely, lower scores indicate weaker beliefs.

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University Health Services Vocational School, Department of Health Care Services Elderly Care, Antalya, Türkiye, Antalya, Konyaaltı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No